CLINICAL TRIAL: NCT04618159
Title: Does Helipyl Eradicate
Acronym: Helipyl
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Yvan Vandenplas, head of departement, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-380
Record Dates: First submitted 2018-10-08; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Eradication

STUDY DESIGN:
Intervention Model Description: helipyl is given to patients with non symptomatic helicobacter pylori infection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Helipyl (Other): helipyl wil be given to 10 children with asymptomatical helicobacter pylori infection
  Interventions: Other: lactobacillus reuteri DSMZ 17648

INTERVENTIONS:
Other: lactobacillus reuteri DSMZ 17648 — to evaluate if this product can eradicate helicobacter pylori

SUMMARY:
Helipyl is on the market; actually it is a post-biotic because it is a killed Lactobacillus reuteri DSMZ 17648. The aim is to demonstrate (or not) that this product eradicates helicobacter, which it claims to do.

DETAILED DESCRIPTION:
This is a pilot project. There is quite limited literature on this product and Helicobacter pylori eradication. My personal opinion is that the literature and guidelines are contradictory. The European guideline is that Helicobacter pylori should not be corrected unless there are "serious" symptoms . On the other hand, Helicobacter is a carcinogen. Quite often, parents ask us, children's gastroenterologists, to screen their children for Helicobacter because they are symptomatic and are being eradicated, and know that Helicobacter is contagious. This creates a difficult situation: not answering the question is not an option according to the parents' opinion. Going into the question and eradicating "classic" is against all guidelines.

Hence this pilot project: 10 complaints-free carriers of Helicobacter pylori (> 5 years) will be treated with Helipyl for one month (product supplied by the company). Beforehand, at the end of the treatment and a month after stopping of the treatment, we do a C13 breath test.

ELIGIBILITY:
Inclusion Criteria:

* >5 and <18 years
* male and female
* asymptomatic helicobacter pylori

Exclusion Criteria:

* helicobacter pylori infection with symptoms
* <5 years

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
to evaluate the C13 breathtest | 6months
  evaluation of C13 breathtest before, at the end of treatment and one month after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Brussel Hoofdstedelijk Gewest, Belgium

IPD SHARING:
Plan to Share IPD: Undecided